CLINICAL TRIAL: NCT04026607
Title: Efficacy of Higher Versus Lower Quality Protein Supplementation to Support Increased Muscle Protein Synthesis in Older Men
Brief Title: Protein Quality to Support Increased Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7360
Record Dates: First submitted 2019-07-15; First posted 2019-07-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Muscle; Aging; Muscle Protein Synthesis
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: The study will be a double blind, randomized parallel group controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and the investigators will be blinded to the supplement type, only the Lead Principal Investigator will have the codes to decipher the supplement type. Supplements are referred to as A, B and C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey Protein Supplement (Experimental): Supplements will be consumed twice daily (25g per serving x 2 servings/day)
  Interventions: Dietary Supplement: Protein Supplementation
- Pea Protein Supplement (Experimental): Supplements will be consumed twice daily (25g per serving x 2 servings/day)
  Interventions: Dietary Supplement: Protein Supplementation
- Collagen Protein Supplement (Experimental): Supplements will be consumed twice daily (25g per serving x 2 servings/day)
  Interventions: Dietary Supplement: Protein Supplementation

INTERVENTIONS:
Dietary Supplement: Protein Supplementation — Participants will continue to ingest the standardized diet; however, supplements will be consumed twice daily (25g per serving x 2 servings/day or 50g supplemental protein/day)

SUMMARY:
The age-related decline in muscle mass and strength is collectively referred to as sarcopenia. Canadian recommended daily allowance (RDA) for protein intake (0.8 g/kg/d), however, many expert groups have advocated that older persons should increase their daily intake to ~1.2 g/kg/d to support the preservation of muscle mass. The use of plant-based proteins in food formulation has recently become of interest. This study will examine the impact of consuming higher- versus lower-quality protein supplements on muscle protein synthesis in healthy older men.

DETAILED DESCRIPTION:
This study will examine the impact of consuming higher- versus lower-quality protein supplements on the integrated rates of muscle protein synthesis in healthy older men. Briefly, participants will consume dietary protein at the RDA for the entire duration of the protocol (2 weeks). Participants will be randomized to consuming collagen (control - CON), whey (WHEY), or pea (PEA) protein supplements twice daily for one week. We will examine the ability of different qualities of protein supplements to stimulate integrated rates of muscle protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Men, between the ages of 65 - 80 years (inclusive)
2. Willing and able to provide informed consent
3. Be in general good health, non-smoking
4. Have a body mass index (BMI) between 20-38 kg/m2 (inclusive)

Exclusion Criteria:

1. Use of tobacco or related products.
2. Veganism or vegetarianism
3. Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements.
4. Use assistive walking devices (e.g., cane or walker)
5. History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
6. Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude oral protein supplement ingestion and/or assessment of safety and study objectives.
7. Any cachexia-related condition (e.g., relating to cancer, tuberculosis or human immunodeficiency virus infection and acquired immune deficiency syndrome) or any genetic muscle diseases or disorders
8. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing)
9. Hypersensitivity or known allergy to any of the components in the test formulations.
10. Excessive alcohol consumption (>21 units/week)
11. History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy (up to 81mg of baby aspirin per day taken as a prophylactic is permitted).
12. History of statin myalgia.
13. Personal or family history of clotting disorder or deep vein thrombosis;
14. Routine/daily usage of non-steroidal anti-inflammatory drugs (NSAIDS, prescription use or daily use of over the counter medication), use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), any anabolic steroid, creatine, whey protein supplements, casein or branched-chain amino acids (BCAAs) within 45 days prior to screening.

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Integrated Muscle Protein Synthesis | 7 days x 2
  Integrated protein synthesis will be determined during 7 days of consuming the RDA of protein (control phase), and during 7 days of supplementation with a randomised protein supplement (Supplement phase).
  Integrated rates of muscle protein synthesis (MPS) will be determined using the D2O method. Briefly, 2H enrichment of saliva (precursor) and muscle (product) pools (relative to 1H) will be determined using isotope ratio mass spectrometry and 'myofibrillar fractional synthetic rate' (%/day) determined.

SECONDARY OUTCOMES:
Anabolic Signalling Proteins | 1 hour
  The effect of each protein supplement on anabolic signalling proteins 1h post-ingestion.
  Briefly, the phosphorylation status (activation) of anabolic signalling proteins will be determined by western blot analysis, and the fold change from that basal state will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University
Locations (1):
- Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKendry J, Lowisz CV, Nanthakumar A, MacDonald M, Lim C, Currier BS, Phillips SM. The effects of whey, pea, and collagen protein supplementation beyond the recommended dietary allowance on integrated myofibrillar protein synthetic rates in older males: a randomized controlled trial. Am J Clin Nutr. 2024 Jul;120(1):34-46. doi: 10.1016/j.ajcnut.2024.05.009. Epub 2024 May 16. PMID 38762187